CLINICAL TRIAL: NCT05782452
Title: Genetic Diagnosis and Phenotype-genotype Correlation in a Large Chinese Cohort of Congenital Cataracts
Brief Title: Genetic Diagnosis in Congenital Cataracts
Status: Completed | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Weirong Chen, Prof., Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2020KYPJ004
Record Dates: First submitted 2023-03-12; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Congenital Cataract
Keywords: Congenital cataract; Genetic diagnosis; Phenotype-genotype correlation
MeSH Terms: interventions — Exome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bilateral congenital cataract probands who were consecutively enrolled
  Interventions: Procedure: Ophthalmic examination; Genetic: Whole-exome sequencing

INTERVENTIONS:
Procedure: Ophthalmic examination — Facial photographs of the participants were obtained at the time of enrolment. Pre- and post-operative anterior eye segment photographs were obtained under diffuse, direct focal and retro illumination. Clinical data, including basic information, family history, and comprehensive pre- and post-operative ophthalmic examination findings, were recorded.
Genetic: Whole-exome sequencing — Performing whole-exome sequencing and bioinformatics analysis.

SUMMARY:
The prediction of genetic risk in congenital cataract patients has great clinical significance. In this trial, the investigators aim to screen the causative variants from 115 unrelated bilateral congenital cataract patients enrolled consecutively, describe novel and recurrent variants, analyze the factors affecting genetic diagnostic yield, and explore potential phenotype-genotype correlation.

DETAILED DESCRIPTION:
Determining whether the disease is hereditary and the precise genetic cause of congenital cataract has great clinical significance in guiding genetic counseling and improving clinical care pathway. Varying among studies, genetic causes account for 8.3-85% of congenital cataracts because of the difference in ethnic background, genetic screening techniques used, the percentage of patients with bilateral cataracts, with a family history, and with syndromic disease.

A phenotype-genotype correlation may be used to predict the causative genes, and the involvement of other tissues and organs based on the appearance of the lens. In addition, it can be used to improve our understanding of lens biology. A phenotype-genotype correlation is difficult to establish because of the genotypic and phenotypic heterogeneity of congenital cataracts.

In this trail, the investigators aim to screen the causative variants from 115 unrelated bilateral congenital cataract patients enrolled consecutively, describe novel and recurrent variants, analyze the factors affecting genetic diagnostic yield, and explore potential phenotype-genotype correlation. Facial and anterior eye segment photographs, pre- and post-operative ocular parameters, and medical and family histories were recorded. Bioinformatics analysis was performed using whole-exome sequencing data. Statistical and correlation analyses were performed using the basic characteristics, deep phenotype, and genotype data.

ELIGIBILITY:
Inclusion Criteria:

1. The participant with bilateral congenital cataract;
2. Have signed a consent form. .

Exclusion Criteria:

1. The participant not identified with congenital cataract; 2. The participant with unilateral congenital cataract.

-

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: This prospective study was a part of an ongoing series at the Childhood Cataract Program of the Chinese Ministry of Health (CCPMOH), China. The cohort consisted of 115 bilateral congenital cataract probands who were consecutively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Whether the participant has pathogenic genes | 2 years
Type of the cataracts | before surgery
  The cataracts were categorized into 17 groups (Membranous cataract, Thin and fibrotic nuclear cataract, Nuclear cataract, Zonular cataract, Pulverulent cataract, Pocket-like cataract, "Ant egg" cataract, Cerulean cataract, Coronary cataract, Coralliform cataract, Cortical cataract, Sutural cataract, Anterior subcapsular cataract, Anterior polar cataract, Posterior subcapsular cataract, Posterior polar cataract, Total cataract)

SECONDARY OUTCOMES:
Whether the participant has family history | 2 years
The symmetricity of the type of cataract | before surgery

CONTACTS AND LOCATIONS:
Overall Officials: Weirong Chen, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Shiels A, Hejtmancik JF. Biology of Inherited Cataracts and Opportunities for Treatment. Annu Rev Vis Sci. 2019 Sep 15;5:123-149. doi: 10.1146/annurev-vision-091517-034346. PMID 31525139
- [Result] Haargaard B, Wohlfahrt J, Fledelius HC, Rosenberg T, Melbye M. Incidence and cumulative risk of childhood cataract in a cohort of 2.6 million Danish children. Invest Ophthalmol Vis Sci. 2004 May;45(5):1316-20. doi: 10.1167/iovs.03-0635. PMID 15111583
- [Result] Gillespie RL, O'Sullivan J, Ashworth J, Bhaskar S, Williams S, Biswas S, Kehdi E, Ramsden SC, Clayton-Smith J, Black GC, Lloyd IC. Personalized diagnosis and management of congenital cataract by next-generation sequencing. Ophthalmology. 2014 Nov;121(11):2124-37.e1-2. doi: 10.1016/j.ophtha.2014.06.006. Epub 2014 Aug 19. PMID 25148791
- [Result] Feinmann J. The BMJ Christmas appeal 2016-17: changing children's lives through cataract surgery. BMJ. 2016 Dec 15;355:i6650. doi: 10.1136/bmj.i6650. No abstract available. PMID 27979852
- [Result] Scott MH, Hejtmancik JF, Wozencraft LA, Reuter LM, Parks MM, Kaiser-Kupfer MI. Autosomal dominant congenital cataract. Interocular phenotypic variability. Ophthalmology. 1994 May;101(5):866-71. doi: 10.1016/s0161-6420(94)31246-2. PMID 8190472
- [Result] Aldahmesh MA, Khan AO, Mohamed JY, Hijazi H, Al-Owain M, Alswaid A, Alkuraya FS. Genomic analysis of pediatric cataract in Saudi Arabia reveals novel candidate disease genes. Genet Med. 2012 Dec;14(12):955-62. doi: 10.1038/gim.2012.86. Epub 2012 Aug 30. PMID 22935719
- [Result] Ng D, Thakker N, Corcoran CM, Donnai D, Perveen R, Schneider A, Hadley DW, Tifft C, Zhang L, Wilkie AO, van der Smagt JJ, Gorlin RJ, Burgess SM, Bardwell VJ, Black GC, Biesecker LG. Oculofaciocardiodental and Lenz microphthalmia syndromes result from distinct classes of mutations in BCOR. Nat Genet. 2004 Apr;36(4):411-6. doi: 10.1038/ng1321. Epub 2004 Mar 7. PMID 15004558
- [Result] Chen J, Ma Z, Jiao X, Fariss R, Kantorow WL, Kantorow M, Pras E, Frydman M, Pras E, Riazuddin S, Riazuddin SA, Hejtmancik JF. Mutations in FYCO1 cause autosomal-recessive congenital cataracts. Am J Hum Genet. 2011 Jun 10;88(6):827-838. doi: 10.1016/j.ajhg.2011.05.008. PMID 21636066
- [Result] Musleh M, Hall G, Lloyd IC, Gillespie RL, Waller S, Douzgou S, Clayton-Smith J, Kehdi E, Black GC, Ashworth J. Diagnosing the cause of bilateral paediatric cataracts: comparison of standard testing with a next-generation sequencing approach. Eye (Lond). 2016 Sep;30(9):1175-81. doi: 10.1038/eye.2016.105. Epub 2016 Jun 17. PMID 27315345
- [Result] Rechsteiner D, Issler L, Koller S, Lang E, Bahr L, Feil S, Ruegger CM, Kottke R, Toelle SP, Zweifel N, Steindl K, Joset P, Zweier M, Suter AA, Gogoll L, Haas C, Berger W, Gerth-Kahlert C. Genetic Analysis in a Swiss Cohort of Bilateral Congenital Cataract. JAMA Ophthalmol. 2021 Jul 1;139(7):691-700. doi: 10.1001/jamaophthalmol.2021.0385. PMID 34014271
- [Result] Kandaswamy DK, Prakash MVS, Graw J, Koller S, Magyar I, Tiwari A, Berger W, Santhiya ST. Application of WES Towards Molecular Investigation of Congenital Cataracts: Identification of Novel Alleles and Genes in a Hospital-Based Cohort of South India. Int J Mol Sci. 2020 Dec 16;21(24):9569. doi: 10.3390/ijms21249569. PMID 33339270